CLINICAL TRIAL: NCT05244746
Title: Efficacy of Ultrasound Guided Rectus Sheath Block Combined With General Anaesthesia on the Postoperative Quality of Recovery Profile in Laparotomy Surgeries, Randomized Control Trial.
Brief Title: Efficacy of Ultrasound Guided Rectus Sheath Block on Post Operative Quality of Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ayman Abougabal, A abougabal, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MS-202-2021
Record Dates: First submitted 2022-02-11; First posted 2022-02-17 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rectus sheath block (Active Comparator)
  Interventions: Procedure: rectus sheath block
- Control (Placebo Comparator)
  Interventions: Procedure: rectus sheath block

INTERVENTIONS:
Procedure: rectus sheath block — blocking the nerve underneath the rectus muscle by bupivicaine

SUMMARY:
Effective Postoperative pain management following laparotomy represents a cornerstone in the care of surgical patients. With the growing utilization of Enhanced recovery after surgery protocols (ERAS), a paradigm shift in perioperative care has resulted in reduction of both hospital stay and clinical complications faced by patients.

One important component of successful implementation of ERAS protocol is optimized pain control. It has been shown that opioids have a considerable role in reducing bowel motility in addition; it hinders early mobilization and enteral feeding besides their commonly faced side effects such as nausea and vomiting.

Consequently, ERAS programs encourage the usage of multimodal opioid sparing analgesia which includes neuraxial or regional anesthesia techniques to provide effective pain relief while reducing the opioid related side effects. [1]

Regional blocks have remained popular with evidence of superior postoperative pain control when compared with systemic analgesics. Regional anaesthesia techniques have undergone considerable refinement with the advent of ultrasound guidance. Ultrasound visualization of anatomical structures increases both the safety and quality of regional blocks through optimal needle placement. Ultrasound-guided rectus sheath (RS) blocks are an emerging anaesthetic technique providing excellent analgesia after laparotomy. The anatomic characteristics of this block suggest minimal serious complications are likely, and this regional block is particularly useful where epidural is contraindicated

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years old patients
2. ASA 1-2 patients
3. Patients undergoing elective midline laparotomy.

Exclusion Criteria:

* 1. refusal to consent, 2. previous laparotomy (subsequently amended to exclude only a laparotomy with a paramedian scar), 3. significant hepatic or renal disease, 4. any condition limiting the use of co-analgesics (diclofenac and acetaminophen), 5. coagulopathy (international normalized ratio: 1.5 ) 6. Patients with body weight \ 50 kg.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
quality of recovery | 24 hours
  using QOR-15 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes